CLINICAL TRIAL: NCT04568863
Title: A Phase II, Single-center, Double-blind, Randomized Placebo-controlled Trial to Explore the Efficacy and Safety of Intravenous Melatonin in Patients With COVID-19 Admitted to the Intensive Care Unit (MelCOVID Study)
Brief Title: Efficacy of Intravenous Melatonin on Mortality in Adult Patients Admitted to the Intensive Care Unit With COVID-19
Acronym: MELCOVID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pharmamel S.L. (Industry)
Collaborators: Hospital Universitario La Paz (Other); Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PHM-2020-001
Record Dates: First submitted 2020-09-28; First posted 2020-09-29 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2020-09

CONDITIONS: COVID-19; SARS-CoV 2; Coronavirus Infection
Keywords: Melatonin intravenous; Placebo intravenous; ICU patients; COVID-19
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Intervention Model Description: phase II, single-center, double-blind, randomized placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin (Experimental): (12 patients): 7 days of 5 mg per Kg of actual body weight per day of intravenous melatonin every 6 hours. Maximum daily dose 500 mg per day.
  Interventions: Drug: Melatonin intravenous
- Placebo (Placebo Comparator): (6 patients): 7 days of 5 mg per Kg of actual body weight per day of intravenous identically-looking placebo every 6 hours.
  Interventions: Drug: Placebo intravenous

INTERVENTIONS:
Drug: Melatonin intravenous — 7 days of 5 mg per Kg of actual body weight per day of intravenous melatonin every 6 hours. Maximum daily dose 500 mg per day.
  Arms: Melatonin
Drug: Placebo intravenous — 7 days of 5 mg per Kg of actual body weight per day of intravenous identically-looking placebo every 6 hours.
  Arms: Placebo

SUMMARY:
There is an urgent need to evaluate effective treatments for COVID-19 patients. Melatonin has significant anti-inflammatory and antioxidant properties and it lacks of side-effects. This randomized controlled trial seeks to evaluate the efficacy of intravenous melatonin in reducing mortality in Covid-19 patients in the ICUs.

DETAILED DESCRIPTION:
ICU COVID-19 patients show high risk of death mainly due to sepsis and respiratory disfunction. Prevention of these critical conditions is mandatory to reduce mortality and to improve patient's outcome.

Melatonin is an endogenous hormone involved not only in circadian rhythm control, but also in the cell protection due to its outstanding anti-inflammatory and antioxidative effects. High doses of melatonin have shown high efficacy against bacterial (sepsis) and viral infections. Melatonin is a safe product that consistently has shown lack of side-effects when it is administered to humans.

SARS-CoV 2 infection may yield severe forms of the disease that require the patients admission to the ICU. These patients may develop an excessive inflammatory response and a burst of free radicals, constituting the major cause of death in these subjects.

Our hypothesis is that high doses of melatonin intravenously administered to COVID-19 ICU patients might reach enough blood levels able to prevent/counteract the developing of sepsis and the production of free radicals, reducing mortality and hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Patient, family member or legal guardian has provided written Informed Consent.
* Age ε 18 years.
* Confirmed SARS-CoV-2 infection with compatible symptoms AND a positive RT-PCR.
* Admission to the ICU with acute hypoxemic respiratory failure attributed to SARS-CoV-2 infection.
* ICU length of stay of less than 7 days prior to randomization with or without MV and without signs of improvement in respiratory failure (MURRAY score at randomization greater or equal to the MURRAY score at ICU admission).

Exclusion Criteria:

* Participant in a different COVID-19 study in which the study drug is under clinical development and hasn't been previously authorized for commercialization.
* Liver enzymes > 5 times the upper normal range.
* Chronic kidney disease with GFR < 30 mL/min/1.73 m2 (stage 4 or greater) or need for hemodialysis.
* Pregnancy. A pregnancy test will be performed on every woman younger than 55 years of age prior to inclusion.
* Terminal surgical or medical illness.
* Autoimmune disease.
* Any patient condition that can prevent the study procedures to be carried out at the treating physician's judgement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-06-20 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Mortality | one month
  Mortality in each study group represented in frequency and time-to-event at day 28 after randomization

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario La Paz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rodriguez-Rubio M, Figueira JC, Acuna-Castroviejo D, Borobia AM, Escames G, de la Oliva P. A phase II, single-center, double-blind, randomized placebo-controlled trial to explore the efficacy and safety of intravenous melatonin in patients with COVID-19 admitted to the intensive care unit (MelCOVID study): a structured summary of a study protocol for a randomized controlled trial. Trials. 2020 Aug 5;21(1):699. doi: 10.1186/s13063-020-04632-4. PMID 32758298
- [Background] Acuna-Castroviejo D, Escames G, Figueira JC, de la Oliva P, Borobia AM, Acuna-Fernandez C. Clinical trial to test the efficacy of melatonin in COVID-19. J Pineal Res. 2020 Oct;69(3):e12683. doi: 10.1111/jpi.12683. Epub 2020 Aug 8. PMID 32770854